CLINICAL TRIAL: NCT00010907
Title: Preliminary Human Trial of NPI-028
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: P50AT000009-02P1 (NIH); 5-P50AT00009-3
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism

INTERVENTIONS:
Drug: NPI-028

SUMMARY:
This research will determine whether the Chinese herbal medicine (NPI-028) can make a significant contribution to the management of withdrawal and to follow-up treatment aimed at preventing or managing relapse in both women and men alcoholics. The herbal preparation has been used historically in the treatment of alcohol intoxication and is still prescribed in China and Southeast Asia. Efficacy has been documented but awaits the application of current research methods to establish efficacy, safety, and probable mechanisms of action. Preclinical studies have been carried out in alcohol-preferring rats and vervet monkeys to test efficacy in reducing voluntary alcohol intake, measure tolerance effects, and toxicological affects. The proposed human trial will develop a placebo, establish quality control, test methods of administration, and examine compliance issues. Following these preliminary steps, a placebo controlled trial will be conducted using 160 subjects (80 subjects per treatment condition with 40 of each gender). Alcohol use, craving, health status, psychological status, and at rates will be assessed using established measures that are current in addiction research.

ELIGIBILITY:
Inclusion Criteria:

* Able to participate as an outpatient
* Considered of acceptable health as determined by physical examination
* English speaking/reading
* Meets DSM-IV criteria for Alcohol Dependence
* Have at least 10 drinking days in the past month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milton L. Bullock, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis